CLINICAL TRIAL: NCT03318523
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study, With an Active-Treatment Dose-Blinded Period, to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of BIIB054 in Subjects With Parkinson's Disease
Brief Title: Evaluating the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of BIIB054 in Participants With Parkinson's Disease
Acronym: SPARK
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: SPARK did not meet it's primary outcome measure for year 1 and failed to meet secondary outcome measures resulting in the development of BIIB054 (cinpanemab) for Parkinson's disease to be discontinued and SPARK study was closed.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 228PD201; 2016-004610-95 (EudraCT Number)
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Results first posted 2021-11-23 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Parkinson's Disease
Keywords: BIIB054; Alpha-synuclein
MeSH Terms: conditions — Parkinson Disease; Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Year 1: Participants will receive matching placebo to BIIB054 on Day 1 and then every 4 weeks.
  Year 2: Participants who received placebo in year 1 will be randomized into one of the active treatment arms in year 2 and will receive BIIB054 intravenous (IV) infusion on Week 52 and then every 4 weeks.
  Interventions: Drug: Placebo
- BIIB054 250 mg (Experimental): Participants will receive BIIB054 250 milligrams (mg) intravenous (IV) infusion on Day 1 and then every 4 weeks.
  Interventions: Drug: BIIB054
- BIIB054 1250 mg (Experimental): Participants will receive BIIB054 1250 mg IV infusion on Day 1 and then every 4 weeks.
  Interventions: Drug: BIIB054
- BIIB054 3500 mg (Experimental): Participants will receive BIIB054 3500 mg IV infusion on Day 1 and then every 4 weeks.
  Interventions: Drug: BIIB054

INTERVENTIONS:
Drug: Placebo — Administered as specified in the treatment arm
  Arms: Placebo
Drug: BIIB054 — Administered as specified in the treatment arm.
  Arms: BIIB054 1250 mg; BIIB054 250 mg; BIIB054 3500 mg

SUMMARY:
The primary objective of the study is to evaluate the clinical efficacy of BIIB054 via dose response using the change from baseline in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Total Score.

The secondary objectives of the study are to evaluate the dose-related safety of BIIB054, to evaluate the clinical efficacy of BIIB054 via MDS-UPDRS total score, to assess the pharmacokinetic (PK) profile of BIIB054, to evaluate the clinical efficacy of BIIB054 based on MDS-UPDRS subparts, to evaluate the pharmacodynamic effects of BIIB054 on the integrity of nigrostriatal dopaminergic nerve terminals and to evaluate the immunogenicity of BIIB054.

ELIGIBILITY:
Inclusion Criteria

* Diagnosed with Parkinson's disease (PD) within a maximum of 3 years prior to Screening.
* Score of ≤2.5 on the Modified Hoehn and Yahr Scale.
* Has not received any medication for the treatment of the motor symptoms of PD for at least 12 weeks prior to Day 1 and, in the opinion of the Investigator, is not expected to require PD treatment for at least 6 months following Day 1. Maximum total duration of prior PD regimens should not exceed 30 days. Stable (at least 8 weeks) dosages of medications that are used to treat conditions other than PD tremor are allowed. Further guidance will be provided by the study's Medical Monitor on a case by case basis.
* Screening dopamine transporter (DaT)/ single-photon emission computed tomography (SPECT) results consistent with neurodegenerative Parkinsonism (central reading).
* All women of childbearing potential and all men must practice highly effective contraception during the study and for 6 months after their last dose of study treatment.

Exclusion Criteria:

* Presence of freezing of gait.
* Montreal cognitive assessment (MOCA) score <23 or other significant cognitive impairment or clinical dementia that, in the opinion of the Investigator, would interfere with study evaluation.
* History of or screening brain magnetic resonance imaging (MRI) scan indicative of clinically significant abnormality, as read by central reader.
* History of severe allergic or anaphylactic reactions, or history of hypersensitivity to BIIB054 or any of the inactive ingredients in the drug product or to radioligands or iodine used in the study.
* Participation in any active immunotherapy study targeting alpha-synuclein.
* Use of allowed medications not previously specified at doses that have not been stable for at least 8 weeks before Day 1, and/or that are not expected to remain stable for the duration of the study.
* Clinically significant abnormal laboratory test values at Screening, as determined by the Investigator.
* Blood donation (1 unit or more) within 8 weeks before Day 1 (must also refrain from donating blood for the duration of the study).

NOTE : Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2021-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (72):
- United States (32):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - St. Joseph's Hopsital & Medical Center- Barrow Neurological Institute, Phoenix, Arizona
  - Research Site, La Jolla, California
  - Cedars Sinai, Los Angeles, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Research Site, Stanford, California
  - University of Colorado Health, Aurora, Colorado
  - Rocky Mountain Movement Disorders Center, PC, Englewood, Colorado
  - Parkinson's Disease and Movement Disorders Centerf, Boca Raton, Florida
  - Mayo Clinic Hospital, Jacksonville, Florida
  - Bioclinica Research, Orlando, Florida
  - USF Health Byrd Institute, Tampa, Florida
  - Northwestern University PD and Movement Disorders Center, Chicago, Illinois
  - Research Site, Chicago, Illinois
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Ochsner Health System, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - NYU Langone Health Center, New York, New York
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Booth Gardner Parkinson's Care Center at Evergreen Health, Kirkland, Washington
  - Inland Northwest Research, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Research Site, Innsbruck, Austria
- Canada (2):
  - University Health Network, Toronto, Ontario
  - Montreal Neurological Institute Clinical Research Unit, Montreal, Quebec
- France (5):
  - Research Name, Toulouse, Haute Garonne
  - CHU Nantes - Hopital Nord Laënnec, Nantes, Loire Atlantique
  - Hopital Roger Salengro - CHU Lille, Lille, Nord
  - Hôpital Henri Mondor, Créteil, Val De Marne
  - Research Site, Paris
- Germany (6):
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum rechts der Isar der TU Muenchen, Munich, Bavaria
  - Universitaetsklinikum Wuerzburg, Würzburg, Bavaria
  - Paracelsus-Elena-Klinik, Kassel, Hesse
  - Universitaetsklinikum Aachen AOeR, Aachen, North Rhine-Westphalia
  - Research Site, Bochum, North Rhine-Westphalia
- Israel (2):
  - Research Site, Haifa
  - Research Site, Tel Aviv
- Italy (10):
  - I.R.C.C.S. Neuromed-Istituto Neurologico Mediterraneo, Pozzilli, Isernia
  - Ospedale Bellaria, Bologna
  - Azienda Ospedaliero Univ. Policlinico Gaspare Rodolico, Catania
  - Research Site, Milan
  - Ospedale San Raffaele, Milan
  - Seconda Università degli Studi di Napoli, Napoli
  - Research Site, Pisa
  - IRCCS San Raffaele, Roma
  - Azienda Ospedaliera Universitaria OO. RR. S. Giovanni di Dio e Ruggi D'Aragona, Salerno
  - Azienda Ospedaliera Santa Maria di Terni, Terni
- Spain (8):
  - Hospital General de Catalunya, Sant Cugat Del Vallés, Barcelona
  - Research Site, Móstoles, Madrid
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Biocruces Health Research Institute, Barakaldo, Vizcaya
  - Hospital Clinic De Barcalona, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Research Site, Madrid
  - Research Site, Seville
- United Kingdom (6):
  - Research Site, Cambridge, Cambridgeshire
  - Salford Royal, Salford, Greater Manchester
  - Research Site, Oxford, Oxfordshire
  - Clinical Ageing Research Unit, Newcastle upon Tyne, Tyne & Wear
  - Royal Hallamshire Hospital, Sheffield, West Midlands
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on http://clinicalresearch.biogen.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Hutchison RM, Fraser K, Yang M, Fox T, Hirschhorn E, Njingti E, Scott D, Bedell BJ, Kistner KM, Cedarbaum JM, Evans KC, Graham D, Martarello L, Mollenhauer B, Lang AE, Dam T, Beaver J. Cinpanemab in Early Parkinson Disease: Evaluation of Biomarker Results From the Phase 2 SPARK Clinical Trial. Neurology. 2024 Mar 12;102(5):e209137. doi: 10.1212/WNL.0000000000209137. Epub 2024 Feb 5. PMID 38315945
- [Derived] Lang AE, Siderowf AD, Macklin EA, Poewe W, Brooks DJ, Fernandez HH, Rascol O, Giladi N, Stocchi F, Tanner CM, Postuma RB, Simon DK, Tolosa E, Mollenhauer B, Cedarbaum JM, Fraser K, Xiao J, Evans KC, Graham DL, Sapir I, Inra J, Hutchison RM, Yang M, Fox T, Budd Haeberlein S, Dam T; SPARK Investigators. Trial of Cinpanemab in Early Parkinson's Disease. N Engl J Med. 2022 Aug 4;387(5):408-420. doi: 10.1056/NEJMoa2203395. PMID 35921450
- [Derived] Hutchison RM, Evans KC, Fox T, Yang M, Barakos J, Bedell BJ, Cedarbaum JM, Brys M, Siderowf A, Lang AE. Evaluating dopamine transporter imaging as an enrichment biomarker in a phase 2 Parkinson's disease trial. BMC Neurol. 2021 Nov 23;21(1):459. doi: 10.1186/s12883-021-02470-8. PMID 34814867
- See also: Fox Trial Finder — https://foxtrialfinder.michaeljfox.org/trial/5100/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 75 investigational sites from 10 January 2018 to 29 April 2021.
Pre-assignment Details: Participants with Parkinson's Disease (PD) were enrolled and randomized to receive placebo or BIIB054 250/1250/3500 milligrams (mg) for Year 1 in Placebo-Controlled (PC) Period. Following Year 1, participants on placebo (delayed start) were re-randomized to receive BIIB054 250/1250/3500 mg dose, and others on BIIB054 in Year 1 continued to receive the same dose until their Week 96 visit.
Groups:
- PC Period: Placebo: Participants received BIIB054-matching placebo, intravenous (IV) infusion, on Day 1 and then every 4 weeks for Year 1 in the PC Period.
- PC Period: BIIB054 250 mg (Early Start): Participants received BIIB054, 250 mg, IV infusion, on Day 1 and then every 4 weeks for Year 1 in the PC Period.
- PC Period: BIIB054 1250 mg (Early Start): Participants received BIIB054, 1250 mg, IV infusion, on Day 1 and then every 4 weeks for Year 1 in the PC Period.
- PC Period: BIIB054 3500 mg (Early Start): Participants received BIIB054, 3500 mg, IV infusion, on Day 1 and then every 4 weeks for Year 1 in the PC Period.
- DBE Period: Placebo to BIIB054 250 mg (Delayed Start): Participants received BIIB054 250 mg, IV infusion from Year 2 up to EOS (approximately 3 years) in the DBE Period. Participants who received placebo in the PC period were included in this arm.
- DBE Period: Placebo to BIIB054 1250 mg (Delayed Start): Participants received BIIB054 1250 mg, IV infusion from Year 2 up to EOS (approximately 3 years) in the DBE Period. Participants who received placebo in the PC period were included in this arm.
- DBE Period: Placebo to BIIB054 3500 mg (Delayed Start): Participants received BIIB054 3500 mg, IV infusion from Year 2 up to EOS (approximately 3 years) in the DBE Period. Participants who received placebo in the PC period were included in this arm.
- DBE Period: BIIB054 250 mg (Early Start): Participants received BIIB054 250 mg, IV infusion from Year 2 up to EOS (approximately 3 years) in the DBE Period. Participants who received BIIB054 250 mg in the PC period were included in this arm.
- DBE Period: BIIB054 1250 mg (Early Start): Participants received BIIB054 1250 mg, IV infusion from Year 2 up to EOS (approximately 3 years) in the DBE Period. Participants who received BIIB054 1250 mg in the PC period were included in this arm.
- DBE Period: BIIB054 3500 mg (Early Start): Participants received BIIB054 3500 mg, IV infusion from Year 2 up to EOS (approximately 3 years) in the DBE Period. Participants who received BIIB054 3500 mg in the PC period were included in this arm.
Period: PC Period: Up to Year 1
Arm/Group | PC Period: Placebo | PC Period: BIIB054 250 mg (Early Start) | PC Period: BIIB054 1250 mg (Early Start) | PC Period: BIIB054 3500 mg (Early Start) | DBE Period: Placebo to BIIB054 250 mg (Delayed Start) | DBE Period: Placebo to BIIB054 1250 mg (Delayed Start) | DBE Period: Placebo to BIIB054 3500 mg (Delayed Start) | DBE Period: BIIB054 250 mg (Early Start) | DBE Period: BIIB054 1250 mg (Early Start) | DBE Period: BIIB054 3500 mg (Early Start)
Started | 100 | 55 | 102 | 100 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 96 | 53 | 100 | 96 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Consent Withdrawn | 3 | 2 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Period: DBE Period:Year 2 to EOS (Up to 3 Years)
Arm/Group | PC Period: Placebo | PC Period: BIIB054 250 mg (Early Start) | PC Period: BIIB054 1250 mg (Early Start) | PC Period: BIIB054 3500 mg (Early Start) | DBE Period: Placebo to BIIB054 250 mg (Delayed Start) | DBE Period: Placebo to BIIB054 1250 mg (Delayed Start) | DBE Period: Placebo to BIIB054 3500 mg (Delayed Start) | DBE Period: BIIB054 250 mg (Early Start) | DBE Period: BIIB054 1250 mg (Early Start) | DBE Period: BIIB054 3500 mg (Early Start)
Started (Out of 345 participants who completed the PC Period, only 344 entered the DBE Period.) | 0 | 0 | 0 | 0 | 20 | 37 | 39 | 52 | 100 | 96
Number of Participants Dosed | 0 | 0 | 0 | 0 | 20 | 37 | 39 | 52 | 100 | 94
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 20 | 37 | 39 | 52 | 100 | 96
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Not completed — Consent Withdrawn | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 2
Not completed — Investigator Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 17 | 36 | 39 | 48 | 94 | 91
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population was defined as all randomized participants who received at least one dose of study treatment (BIIB054 or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | PC Period: Placebo | PC Period: BIIB054 250 mg (Early Start) | PC Period: BIIB054 1250 mg (Early Start) | PC Period: BIIB054 3500 mg (Early Start) | Total
Number analyzed (Participants) | 100 | 55 | 102 | 100 | 357
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (8.39) | 61.3 (9.24) | 59.2 (8.48) | 59.3 (9.92) | 60.1 (9.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 16 | 29 | 34 | 107
  Male | 72 | 39 | 73 | 66 | 250
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 1 | 6 | 11
  Not Hispanic or Latino | 96 | 54 | 101 | 94 | 345
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 2 | 2
  Asian | 0 | 0 | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 96 | 53 | 92 | 84 | 325
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6 | 11 | 23
Baseline Movement Disorder Society Sponsored Revision of the Unified PD Rating Scale Total Score [Mean (Standard Deviation); unit: score on a scale] — Movement Disorder Society Sponsored Revision of the Unified PD Rating Scale (MDS-UPDRS) is multimodal scale assessing impairment and disability consisting of 4 parts. Part I: non-motor experiences of daily living and has 2 components (13 questions[Q], Range[R] 0-52). Part II: motor experiences of daily living (13 Q, R 0-52). Part III: motor signs of PD and was administered by rater (33 Q, R 0-132). Numeric score for each question is between 0-4; 0=Normal,1=Slight,2=Mild,3=Moderate,4=Severe. MDS-UPDRS Total Score=sum of Parts I, II, and III (R 0-236). Higher score=more severe symptoms of PD.
  score on a scale | 31.9 (12.41) | 31.9 (12.25) | 32.9 (12.58) | 32.6 (13.46) | 32.4 (12.69)
Baseline MDS-UPDRS Subpart I Score [Mean (Standard Deviation); unit: score on a scale] — MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. It is separated into 4 subscales: Part I assessed non-motor experiences of daily living and has 2 components (Range 0-52). Part IA contained 6 questions and were assessed by the examiner (Range 0-24). Part IB contained 7 questions on non-motor experiences of daily living which were completed by the participant (Range 0-28). For each question a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. A higher score indicated more severe symptoms of PD.
  score on a scale | 4.3 (3.50) | 3.3 (2.74) | 4.8 (3.99) | 4.3 (3.60) | 4.3 (3.59)
Baseline MDS-UPDRS Subpart II Score [Mean (Standard Deviation); unit: score on a scale] — MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. Part II assessed motor experiences of daily living (Range 0-52). It contained 13 questions completed by the participant. For each question a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. A higher score indicated more severe symptoms of PD.
  score on a scale | 5.4 (3.87) | 5.0 (3.30) | 5.3 (3.66) | 5.5 (4.30) | 5.3 (3.84)
Baseline MDS-UPDRS Subpart III Score [Mean (Standard Deviation); unit: score on a scale] — MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. Part III assessed the motor signs of Parkinson's Disease (PD) and was administered by the rater (Range 0-132). Part III contained 33 scores based on 18 items. For each question a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. A higher score indicated more severe symptoms of PD.
  score on a scale | 22.2 (9.31) | 23.5 (9.38) | 22.8 (8.69) | 22.9 (8.86) | 22.8 (8.99)
Baseline Total Striatum Striatal Binding Ratio (SBR) [Mean (Standard Deviation); unit: striatal binding ratio] — Population: ITT population. Number analyzed is the number of participants analyzed for this study specific baseline measure.
  striatal binding ratio
    number analyzed (Participants) | 100 | 55 | 102 | 99 | 356
    (all) | 1.295 (0.3177) | 1.409 (0.3875) | 1.342 (0.3197) | 1.351 (0.3495) | 1.342 (0.3393)
Baseline Total Putamen SBR [Mean (Standard Deviation); unit: striatal binding ratio] — Population: ITT population. Number analyzed is the number of participants analyzed for this study specific baseline measure.
  striatal binding ratio
    number analyzed (Participants) | 100 | 55 | 102 | 99 | 356
    (all) | 1.255 (0.3429) | 1.388 (0.4294) | 1.291 (0.3269) | 1.286 (0.3627) | 1.295 (0.3597)
Baseline Total Caudate SBR [Mean (Standard Deviation); unit: striatal binding ratio] — Population: ITT population. Number analyzed is the number of participants analyzed for this study specific baseline measure.
  striatal binding ratio
    number analyzed (Participants) | 100 | 55 | 102 | 99 | 356
    (all) | 1.336 (0.3279) | 1.433 (0.3751) | 1.397 (0.3417) | 1.416 (0.3643) | 1.391 (0.3501)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Movement Disorder Society Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Total Score (Sum of Parts I, II, and III) at Week 52
Description: MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. Part I assessed non-motor experiences of daily living and has 2 components (Range 0-52). Part IA contained 6 questions and were assessed by the examiner (Range 0-24). Part IB contained 7 questions on non-motor experiences of daily living which were completed by the participant (Range 0-28). Part II assessed motor experiences of daily living (Range 0-52). It contained 13 questions completed by the participant. Part III assessed the motor signs of PD and was administered by the rater (Range 0-132). Part III contained 33 scores based on 18 items. For each question a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. MDS-UPDRS Total Score equals the sum of Parts I, II, and III (Range 0-236). A higher score indicated more severe symptoms of PD. The mean values reported are the adjusted mean values.
Time Frame: Baseline, Week 52
Population: The ITT population was defined as all randomized participants who received at least one dose of study treatment (BIIB054 or placebo). Number of participants analyzed were participants analyzed for this outcome measure.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- PC Period: Placebo: Participants received BIIB054-matching placebo, IV infusion, on Day 1 and then every 4 weeks for Year 1 in the PC Period.
- PC Period: BIIB054 1250 mg (Early Start): Participants received BIIB054, 1250 mg, IV infusion, on Day 1 and then every 4 weeks for Year 1 in PC Period.
- PC Period: BIIB054 3500 mg (Early Start): Participants received BIIB054, 3500 mg, IV infusion, on Day 1 and then every 4 weeks for Year 1 in PC Period.
Arm/Group | PC Period: Placebo | PC Period: BIIB054 250 mg (Early Start) | PC Period: BIIB054 1250 mg (Early Start) | PC Period: BIIB054 3500 mg (Early Start)
Number analyzed (Participants) | 53 | 29 | 57 | 51
score on a scale | 10.78 (1.490) | 10.48 (1.951) | 11.29 (1.446) | 10.86 (1.518)
Statistical Analysis 1: Comparison: PC Period: Placebo vs PC Period: BIIB054 250 mg (Early Start); Change From Baseline in MDS-UPDRS Total Score at Week 52; Test type: Superiority — Adjusted mean, difference with placebo, 95% confidence interval (CI), and p-value were based on a mixed model for repeated measures (MMRM) model, with change from baseline in MDS-UPDRS score as dependent variable and with fixed effects of treatment group, time, treatment group-by-time interaction, region, PD subtype, prior use of PD medication, baseline MDS-UPDRS score, baseline MDS-UPDRS by time interaction, baseline striatum SBR values and baseline striatum SBR value by time interaction; p = 0.8976, Mixed Model for Repeated Measures; Difference = -0.30, 95% CI 2-sided [-4.888 to 4.287]
Statistical Analysis 2: Comparison: PC Period: Placebo vs PC Period: BIIB054 1250 mg (Early Start); Change From Baseline in MDS-UPDRS Total Score at Week 52; Test type: Superiority — Adjusted mean, difference with placebo, 95% CI, and p-value were based on an MMRM model, with change from baseline in MDS-UPDRS score as dependent variable and with fixed effects of treatment group, time, treatment group-by-time interaction, region, PD subtype, prior use of PD medication, baseline MDS-UPDRS score, baseline MDS-UPDRS by time interaction, baseline striatum SBR values and baseline striatum SBR value by time interaction; p = 0.7960, Mixed Model for Repeated Measures; Difference = 0.50, 95% CI 2-sided [-3.310 to 4.312]
Statistical Analysis 3: Comparison: PC Period: Placebo vs PC Period: BIIB054 3500 mg (Early Start); Change From Baseline in MDS-UPDRS Total Score at Week 52; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.9695, Mixed Model for Repeated Measures; Difference = 0.08, 95% CI 2-sided [-3.805 to 3.956]

2. Primary Outcome: Change From Baseline in Movement Disorder Society Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Total Score (Sum of Parts I, II, and III) at Week 72
Description: as for outcome 1
Time Frame: Baseline, Week 72
Population: The ITT population was defined as all randomized participants who received at least one dose of study treatment (BIIB054 or placebo). As prespecified in the protocol, the data for the delayed start BIIB054 were pooled from Placebo/BIIB054 250/1250/3500 mg for the analysis of this outcome measure. Number of participants analyzed were participants analyzed for this outcome measure.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled): Participants who received BIIB054-matching placebo in Year 1 followed by BIIB054 250 mg or 1250 mg or 3500 mg, IV infusion from Year 2 up to EOS (approximately 3 years) were pooled in this arm.
- PC Period: Early Start BIIB054 250 mg: Participants received BIIB054, 250 mg, IV infusion, on Day 1 and then every 4 weeks for Year 1 in the PC Period.
- PC Period: Early Start BIIB054 1250 mg: Participants received BIIB054, 1250 mg, IV infusion, on Day 1 and then every 4 weeks for Year 1 in PC Period.
- PC Period: Early Start BIIB054 3500 mg: Participants received BIIB054, 3500 mg, IV infusion, on Day 1 and then every 4 weeks for Year 1 in PC Period.
Arm/Group | PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) | PC Period: Early Start BIIB054 250 mg | PC Period: Early Start BIIB054 1250 mg | PC Period: Early Start BIIB054 3500 mg
Number analyzed (Participants) | 68 | 32 | 62 | 64
score on a scale | 7.11 (1.476) | 6.83 (2.032) | 8.66 (1.496) | 6.94 (1.508)
Statistical Analysis 1: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 250 mg; Change From Baseline in MDS-UPDRS Total Score at Week 72; Test type: Superiority — Adjusted mean, difference with delayed start group, 95% CI, and p-value were based on an MMRM model, with change from baseline in MDS-UPDRS score as dependent variable and with fixed effects of treatment group, time, treatment group-by-time interaction, region, PD subtype, prior use of PD medication, corresponding baseline MDS-UPDRS score, corresponding baseline MDS-UPDRS by time interaction, baseline striatum SBR values and baseline striatum SBR value by time interaction; p = 0.9093, Mixed Model for Repeated Measures; Difference = -0.28, 95% CI 2-sided [-5.035 to 4.483]
Statistical Analysis 2: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 1250 mg; Change From Baseline in MDS-UPDRS Total Score at Week 72; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.4327, Mixed Model for Repeated Measures; Difference = 1.55, 95% CI 2-sided [-2.336 to 5.440]
Statistical Analysis 3: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 3500 mg; Change From Baseline in MDS-UPDRS Total Score at Week 72; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.9330, Mixed Model with repeated Measures; Difference = -0.17, 95% CI 2-sided [-4.051 to 3.719]

3. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose, results in death; in the view of the investigator places the participant at immediate risk of death; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect; is a medically important event.
Time Frame: Up to 3 years
Population: The safety population was defined as all participants who received at least one dose of study treatment (BIIB054).
Measure: Number; unit: percentage of participants
Arm/Group | PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) | PC Period: Early Start BIIB054 250 mg | PC Period: Early Start BIIB054 1250 mg | PC Period: Early Start BIIB054 3500 mg
Number analyzed (Participants) | 96 | 55 | 102 | 100
percentage of participants
  AEs | 77.1 | 85.5 | 89.2 | 93.0
  SAEs | 8.3 | 10.9 | 8.8 | 12.0

4. Secondary Outcome: Change From Baseline in MDS-UPDRS Total Score (Sum of Parts I, II, and III) at Week 96
Description: as for outcome 1
Time Frame: Baseline, Week 96
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) | PC Period: Early Start BIIB054 250 mg | PC Period: Early Start BIIB054 1250 mg | PC Period: Early Start BIIB054 3500 mg
Number analyzed (Participants) | 67 | 28 | 62 | 59
score on a scale | 7.88 (1.616) | 8.28 (2.317) | 8.71 (1.628) | 8.87 (1.659)
Statistical Analysis 1: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 250 mg; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.8828, Mixed Model for Repeated Measures; Difference = 0.41, 95% CI 2-sided [-5.013 to 5.825]
Statistical Analysis 2: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 1250 mg; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.7019, Mixed Model for Repeated Measure; Difference = 0.84, 95% CI 2-sided [-3.458 to 5.128]
Statistical Analysis 3: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 3500 mg; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.6519, Mixed Model for Repeated Measures; Difference = 0.99, 95% CI 2-sided [-3.323 to 5.301]

5. Secondary Outcome: Serum Concentration of BIIB054
Time Frame: Pre-dose and 1 hour post-dose of Baseline, Weeks 4, 8, 12, 16, 24, 32, 36, 44, 52, 60, 68, 84, 96, 120 and 144
Population: The pharmacokinetic (PK) population was defined as all participants in the ITT population who had at least one measurable BIIB054 concentration in serum or cerebrospinal fluid (CSF). Number analyzed is the number of participants analyzed at the specified time point.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (ug/mL)
Groups:
- BIIB054 250 mg: Participants received BIIB054, 250 mg, IV infusion, from Day 1 up to EOS (approximately 3 years).
- BIIB054 1250 mg: Participants received BIIB054, 1250 mg, IV infusion, from Day 1 up to EOS (approximately 3 years).
- BIIB054 3500 mg: Participants received BIIB054, 3500 mg, IV infusion, from Day 1 up to EOS (approximately 3 years).
Arm/Group | BIIB054 250 mg | BIIB054 1250 mg | BIIB054 3500 mg
Number analyzed (Participants) | 75 | 139 | 139
micrograms per milliliter (ug/mL)
  Baseline (Pre-dose): number analyzed (Participants) | 48 | 95 | 92
  Baseline (Pre-dose) | 0.00 (0.000) | 7.47 (51.281) | 0.01 (0.065)
  Baseline (1 Hour Post-dose): number analyzed (Participants) | 62 | 121 | 114
  Baseline (1 Hour Post-dose) | 75.02 (15.829) | 374.79 (86.004) | 1137.28 (335.336)
  Week 4 (Pre-dose): number analyzed (Participants) | 46 | 95 | 91
  Week 4 (Pre-dose) | 20.37 (5.004) | 95.36 (27.882) | 306.20 (95.257)
  Week 4 (1 Hour Post-dose): number analyzed (Participants) | 47 | 94 | 91
  Week 4 (1 Hour Post-dose) | 97.09 (19.711) | 468.56 (190.589) | 1354.19 (364.468)
  Week 8 (Pre-dose): number analyzed (Participants) | 63 | 125 | 122
  Week 8 (Pre-dose) | 29.73 (8.371) | 169.79 (68.025) | 495.79 (153.357)
  Week 8 (1 Hour Post-dose): number analyzed (Participants) | 64 | 127 | 122
  Week 8 (1 Hour Post-dose) | 103.69 (26.964) | 543.91 (143.212) | 1591.57 (465.798)
  Week 12 (Pre-dose): number analyzed (Participants) | 50 | 97 | 96
  Week 12 (Pre-dose) | 36.76 (11.830) | 195.16 (51.020) | 580.43 (185.761)
  Week 12 (1 Hour Post-dose): number analyzed (Participants) | 54 | 99 | 97
  Week 12 (1 Hour Post-dose) | 112.61 (27.378) | 569.41 (141.250) | 1632.29 (459.839)
  Week 16 (Pre-dose): number analyzed (Participants) | 51 | 99 | 98
  Week 16 (Pre-dose) | 40.82 (11.421) | 201.33 (73.451) | 642.06 (194.288)
  Week 16 (1 Hour Post-dose): number analyzed (Participants) | 50 | 99 | 98
  Week 16 (1 Hour Post-dose) | 117.08 (27.401) | 614.85 (186.892) | 1739.98 (506.346)
  Week 24 (Pre-dose): number analyzed (Participants) | 54 | 98 | 94
  Week 24 (Pre-dose) | 43.31 (12.906) | 235.69 (84.454) | 724.60 (228.295)
  Week 24 (1 Hour Post-dose): number analyzed (Participants) | 46 | 90 | 87
  Week 24 (1 Hour Post-dose) | 125.79 (36.695) | 664.26 (209.251) | 1867.92 (470.283)
  Week 32 (Pre-dose): number analyzed (Participants) | 11 | 19 | 24
  Week 32 (Pre-dose) | 42.69 (13.486) | 260.35 (104.397) | 772.75 (299.703)
  Week 32 (1 Hour Post-dose): number analyzed (Participants) | 15 | 25 | 28
  Week 32 (1 Hour Post-dose) | 139.00 (34.758) | 626.16 (164.497) | 1985.71 (497.545)
  Week 36 (Pre-dose): number analyzed (Participants) | 51 | 100 | 96
  Week 36 (Pre-dose) | 45.77 (11.867) | 262.80 (85.052) | 819.83 (328.774)
  Week 36 (1 Hour Post-dose): number analyzed (Participants) | 51 | 100 | 95
  Week 36 (1 Hour Post-dose) | 123.67 (29.536) | 665.60 (145.235) | 1916.84 (543.373)
  Week 44 (Pre-dose): number analyzed (Participants) | 3 | 5 | 7
  Week 44 (Pre-dose) | 58.17 (22.774) | 280.40 (116.590) | 858.43 (349.573)
  Week 44 (1 Hour Post-dose): number analyzed (Participants) | 3 | 5 | 8
  Week 44 (1 Hour Post-dose) | 143.33 (41.004) | 582.40 (194.431) | 2066.25 (579.555)
  Week 52 (Pre-dose): number analyzed (Participants) | 49 | 98 | 82
  Week 52 (Pre-dose) | 46.70 (19.343) | 232.08 (87.529) | 787.35 (341.229)
  Week 52 (1 Hour Post-dose): number analyzed (Participants) | 35 | 74 | 64
  Week 52 (1 Hour Post-dose) | 114.59 (25.913) | 645.36 (264.270) | 1920.78 (479.511)
  Week 60 (Pre-dose): number analyzed (Participants) | 42 | 86 | 84
  Week 60 (Pre-dose) | 43.41 (15.973) | 254.52 (88.446) | 724.77 (314.854)
  Week 60 (1 Hour Post-dose): number analyzed (Participants) | 41 | 83 | 80
  Week 60 (1 Hour Post-dose) | 122.55 (29.374) | 657.94 (149.654) | 1905.43 (494.136)
  Week 68 (Pre-dose): number analyzed (Participants) | 2 | 3 | 2
  Week 68 (Pre-dose) | 706.25 (966.969) | 202.33 (34.210) | 1362.50 (533.866)
  Week 68 (1 Hour Post-dose): number analyzed (Participants) | 2 | 3 | 2
  Week 68 (1 Hour Post-dose) | 171.50 (44.548) | 576.33 (85.290) | 2305.00 (1025.305)
  Week 84 (Pre-dose): number analyzed (Participants) | 28 | 50 | 42
  Week 84 (Pre-dose) | 47.00 (15.535) | 255.54 (81.407) | 746.43 (249.770)
  Week 84 (1 Hour Post-dose): number analyzed (Participants) | 38 | 60 | 52
  Week 84 (1 Hour Post-dose) | 134.91 (33.035) | 648.62 (120.163) | 1942.02 (501.095)
  Week 96 (Pre-dose): number analyzed (Participants) | 11 | 18 | 16
  Week 96 (Pre-dose) | 41.25 (15.345) | 274.56 (71.718) | 654.70 (262.926)
  Week 96 (1 Hour Post-dose): number analyzed (Participants) | 10 | 20 | 16
  Week 96 (1 Hour Post-dose) | 122.00 (29.527) | 682.30 (123.653) | 1822.50 (475.682)
  Week 120 (Pre-dose): number analyzed (Participants) | 6 | 6 | 7
  Week 120 (Pre-dose) | 34.98 (12.042) | 279.00 (99.499) | 727.29 (116.793)
  Week 120 (1 Hour Post-dose): number analyzed (Participants) | 6 | 6 | 7
  Week 120 (1 Hour Post-dose) | 119.67 (15.629) | 769.83 (279.182) | 1717.14 (320.037)
  Week 144 (Pre-dose): number analyzed (Participants) | 0 | 1 | 0
  Week 144 (Pre-dose) |  | 365.00 (NA) — NA: Standard Deviation was not determinable. |
  Week 144 (1 Hour Post-dose): number analyzed (Participants) | 0 | 1 | 0
  Week 144 (1 Hour Post-dose) |  | 721.00 (NA) — NA: Standard Deviation was not determinable. |

6. Secondary Outcome: Change From Baseline in MDS-UPDRS Subpart I Score at Week 52
Description: MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. Part I assessed non-motor experiences of daily living and has 2 components (Range 0-52). Part IA contained 6 questions and were assessed by the examiner (Range 0-24). Part IB contained 7 questions on non-motor experiences of daily living which were completed by the participant (Range 0-28). For each question a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. A higher score indicated more severe symptoms of PD. The mean values reported are the adjusted mean values.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PC Period: Placebo | PC Period: BIIB054 250 mg (Early Start) | PC Period: BIIB054 1250 mg (Early Start) | PC Period: BIIB054 3500 mg (Early Start)
Number analyzed (Participants) | 53 | 29 | 57 | 51
score on a scale | 1.43 (0.436) | 0.90 (0.570) | 1.56 (0.423) | 1.65 (0.446)
Statistical Analysis 1: Comparison: PC Period: Placebo vs PC Period: BIIB054 250 mg (Early Start); Change from Baseline in MDS-UPDRS Subpart I Score at Week 52; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.4327, Mixed Model for Repeated Measures; Difference = -0.53, 95% CI 2-sided [-1.851 to 0.794]
Statistical Analysis 2: Comparison: PC Period: Placebo vs PC Period: BIIB054 1250 mg (Early Start); Change from Baseline in MDS-UPDRS Subpart I Score at Week 52; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.8155, Mixed Model for Repeated Measures; Difference = 0.13, 95% CI 2-sided [-0.965 to 1.225]
Statistical Analysis 3: Comparison: PC Period: Placebo vs PC Period: BIIB054 3500 mg (Early Start); Change from Baseline in MDS-UPDRS Subpart I Score at Week 52; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.7015, Mixed Model for Repeated Measures; Difference = 0.22, 95% CI 2-sided [-0.899 to 1.334]

7. Secondary Outcome: Change From Baseline in MDS-UPDRS Subpart I Score at Weeks 72 and 96
Description: as for outcome 6
Time Frame: Baseline, Weeks 72 and 96
Population: The ITT population was defined as all randomized participants who received at least one dose of study treatment (BIIB054 or placebo). As prespecified in the protocol, the data for the delayed start BIIB054 were pooled from Placebo/BIIB054 250/1250/3500 mg for the analysis of this outcome measure. Number analyzed is the number of participants analyzed at the specified time point.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) | PC Period: Early Start BIIB054 250 mg | PC Period: Early Start BIIB054 1250 mg | PC Period: Early Start BIIB054 3500 mg
Number analyzed (Participants) | 100 | 55 | 102 | 100
score on a scale
  Change from Baseline at Week 72: number analyzed (Participants) | 68 | 32 | 62 | 64
  Change from Baseline at Week 72 | 1.65 (0.395) | 0.61 (0.538) | 1.73 (0.402) | 1.63 (0.405)
  Change from Baseline at Week 96: number analyzed (Participants) | 67 | 28 | 62 | 59
  Change from Baseline at Week 96 | 1.95 (0.398) | 1.69 (0.568) | 1.93 (0.403) | 1.72 (0.414)
Statistical Analysis 1: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 250 mg; Change from Baseline in MDS-UPDRS Subpart I Score at Week 72; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.1038, Mixed Model for Repeated Measures; Difference = -1.03, 95% CI 2-sided [-2.276 to 0.213]
Statistical Analysis 2: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 1250 mg; Change from Baseline in MDS-UPDRS Subpart I Score at Week 72; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.8689, Mixed Model for Repeated Measures; Difference = 0.09, 95% CI 2-sided [-0.933 to 1.103]
Statistical Analysis 3: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 3500 mg; Change from Baseline in MDS-UPDRS Subpart I Score at Week 72; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.9820, Mixed Model for Repeated Measures; Difference = -0.01, 95% CI 2-sided [-1.026 to 1.003]
Statistical Analysis 4: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 250 mg; Change from Baseline in MDS-UPDRS Subpart I Score at Week 96; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.6930, Mixed Model for Repeated Measures; Difference = -0.26, 95% CI 2-sided [-1.563 to 1.040]
Statistical Analysis 5: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 1250 mg; Change from Baseline in MDS-UPDRS Subpart I Score at Week 96; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.9606, Mixed Model for Repeated Measures; Difference = -0.03, 95% CI 2-sided [-1.053 to 1.001]
Statistical Analysis 6: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 3500 mg; Change from Baseline in MDS-UPDRS Subpart I Score at Week 96; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.6512, Mixed Model for Repeated Measures; Difference = -0.24, 95% CI 2-sided [-1.269 to 0.794]

8. Secondary Outcome: Change From Baseline in MDS-UPDRS Subpart II Score at Week 52
Description: MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. Part II assessed motor experiences of daily living (Range 0-52). It contained 13 questions completed by the participant. For each question a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. A higher score indicated more severe symptoms of PD. The mean values reported are the adjusted mean values.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PC Period: Placebo | PC Period: BIIB054 250 mg (Early Start) | PC Period: BIIB054 1250 mg (Early Start) | PC Period: BIIB054 3500 mg (Early Start)
Number analyzed (Participants) | 54 | 29 | 58 | 51
score on a scale | 3.17 (0.473) | 2.72 (0.621) | 3.16 (0.460) | 3.01 (0.486)
Statistical Analysis 1: Comparison: PC Period: Placebo vs PC Period: BIIB054 250 mg (Early Start); Change from Baseline in MDS-UPDRS Subpart II Score at Week 52; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.5497, Mixed Model for Repeated Measures; Difference = -0.44, 95% CI 2-sided [-1.889 to 1.007]
Statistical Analysis 2: Comparison: PC Period: Placebo vs PC Period: BIIB054 1250 mg (Early Start); Change from Baseline in MDS-UPDRS Subpart II Score at Week 52; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.9980, Mixed Model for Repeated Measures; Difference = -0.00, 95% CI 2-sided [-1.200 to 1.197]
Statistical Analysis 3: Comparison: PC Period: Placebo vs PC Period: BIIB054 3500 mg (Early Start); Change from Baseline in MDS-UPDRS Subpart II Score at Week 52; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.8069, Mixed Model for Repeated Measures; Difference = -0.15, 95% CI 2-sided [-1.374 to 1.070]

9. Secondary Outcome: Change From Baseline in MDS-UPDRS Subpart II Score at Weeks 72 and 96
Description: as for outcome 8
Time Frame: Baseline, Weeks 72 and 96
Population: The ITT population was defined as all randomized participants who received at least one dose of study treatment (BIIB054 or placebo). As prespecified in the protocol, the data for the delayed start BIIB054 were pooled from (Placebo/BIIB054 250/1250/3500 mg) for the analysis of this outcome measure. Number analyzed is the number of participants analyzed at the specified time point.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) | PC Period: Early Start BIIB054 250 mg | PC Period: Early Start BIIB054 1250 mg | PC Period: Early Start BIIB054 3500 mg
Number analyzed (Participants) | 100 | 55 | 102 | 100
score on a scale
  Change from Baseline at Week 72: number analyzed (Participants) | 69 | 33 | 62 | 64
  Change from Baseline at Week 72 | 1.83 (0.491) | 1.62 (0.672) | 2.36 (0.497) | 1.68 (0.503)
  Change from Baseline at Week 96: number analyzed (Participants) | 67 | 28 | 62 | 60
  Change from Baseline at Week 96 | 1.87 (0.529) | 1.33 (0.762) | 2.39 (0.533) | 2.22 (0.541)
Statistical Analysis 1: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 250 mg; Change from Baseline in MDS-UPDRS Subpart II Score at Week 72; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.7968, Mixed Model for Repeated Measures; Difference = -0.21, 95% CI 2-sided [-1.786 to 1.372]
Statistical Analysis 2: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 1250 mg; Change from Baseline in MDS-UPDRS Subpart II Score at Week 72; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.4211, Mixed Model for Repeated Measures; Difference = 0.53, 95% CI 2-sided [-0.766 to 1.827]
Statistical Analysis 3: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 3500 mg; Change from Baseline in MDS-UPDRS Subpart II Score at Week 72; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.8166, Mixed Model for Repeated Measures; Difference = -0.15, 95% CI 2-sided [-1.448 to 1.143]
Statistical Analysis 4: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 250 mg; Change from Baseline in MDS-UPDRS Subpart II Score at Week 96; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.5535, Mixed Model for Repeated Measures; Difference = -0.53, 95% CI 2-sided [-2.310 to 1.240]
Statistical Analysis 5: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 1250 mg; Change from Baseline in MDS-UPDRS Subpart II Score at Week 96; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.4654, Mixed Model for Repeated Measures; Difference = 0.52, 95% CI 2-sided [-0.881 to 1.922]
Statistical Analysis 6: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 3500 mg; Change from Baseline in MDS-UPDRS Subpart II Score at Week 96; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.6184, Mixed Model for Repeated Measures; Difference = 0.36, 95% CI 2-sided [-1.051 to 1.763]

10. Secondary Outcome: Change From Baseline in MDS-UPDRS Subpart III Score at Week 52
Description: MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. Part III assessed the motor signs of PD and was administered by the rater (Range 0-132). Part III contained 33 scores based on 18 items. For each question a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. A higher score indicated more severe symptoms of PD. The mean values reported are the adjusted mean values.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PC Period: Placebo | PC Period: BIIB054 250 mg (Early Start) | PC Period: BIIB054 1250 mg (Early Start) | PC Period: BIIB054 3500 mg (Early Start)
Number analyzed (Participants) | 53 | 29 | 58 | 51
score on a scale | 6.10 (1.083) | 6.69 (1.419) | 6.76 (1.046) | 6.20 (1.104)
Statistical Analysis 1: Comparison: PC Period: Placebo vs PC Period: BIIB054 250 mg (Early Start); Change from Baseline in MDS-UPDRS Subpart III Score at Week 52; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.7274, Mixed Model for Repeated Measures; Difference = 0.59, 95% CI 2-sided [-2.742 to 3.925]
Statistical Analysis 2: Comparison: PC Period: Placebo vs PC Period: BIIB054 1250 mg (Early Start); Change from Baseline in MDS-UPDRS Subpart III Score at Week 52; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.6385, Mixed Model for Repeated Measures; Difference = 0.66, 95% CI 2-sided [-2.094 to 3.411]
Statistical Analysis 3: Comparison: PC Period: Placebo vs PC Period: BIIB054 3500 mg (Early Start); Change from Baseline in MDS-UPDRS Subpart III Score at Week 52; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.9467, Mixed Model for Repeated Measures; Difference = 0.10, 95% CI 2-sided [-2.718 to 2.910]

11. Secondary Outcome: Change From Baseline in MDS-UPDRS Subpart III Score at Weeks 72 ad 96
Description: as for outcome 10
Time Frame: Baseline, Weeks 72 and 96
Population: as for outcome 9
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) | PC Period: Early Start BIIB054 250 mg | PC Period: Early Start BIIB054 1250 mg | PC Period: Early Start BIIB054 3500 mg
Number analyzed (Participants) | 100 | 55 | 102 | 100
score on a scale
  Change from Baseline at Week 72: number analyzed (Participants) | 68 | 32 | 62 | 64
  Change from Baseline at Week 72 | 3.64 (1.027) | 4.48 (1.404) | 4.49 (1.038) | 3.69 (1.048)
  Change from Baseline at Week 96: number analyzed (Participants) | 67 | 28 | 62 | 60
  Change from Baseline at Week 96 | 4.49 (1.174) | 5.14 (1.679) | 4.39 (1.180) | 5.17 (1.201)
Statistical Analysis 1: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 250 mg; Change from Baseline in MDS-UPDRS Subpart III Score at Week 72; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.6112, Mixed Model for Repeated Measures; Difference = 0.85, 95% CI 2-sided [-2.423 to 4.114]
Statistical Analysis 2: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 1250 mg; Change from Baseline in MDS-UPDRS Subpart III Score at Week 72; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.5270, Mixed Model for Repeated Measures; Difference = 0.86, 95% CI 2-sided [-1.806 to 3.520]
Statistical Analysis 3: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 3500 mg; Change from Baseline in MDS-UPDRS Subpart III Score at Week 72; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.9673, Mixed Model for Repeated Measures; Difference = 0.06, 95% CI 2-sided [-2.608 to 2.719]
Statistical Analysis 4: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 250 mg; Change from Baseline in MDS-UPDRS Subpart III Score at Week 96; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.7455, Mixed Model for Repeated Measures; Difference = 0.65, 95% CI 2-sided [-3.274 to 4.569]
Statistical Analysis 5: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 1250 mg; Change from Baseline in MDS-UPDRS Subpart III Score at Week 96; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.9506, Mixed Model for Repeated Measures; Difference = -0.10, 95% CI 2-sided [-3.192 to 2.997]
Statistical Analysis 6: Comparison: PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) vs PC Period: Early Start BIIB054 3500 mg; Change from Baseline in MDS-UPDRS Subpart III Score at Week 96; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.6643, Mixed Model for Repeated Measures; Difference = 0.69, 95% CI 2-sided [-2.422 to 3.794]

12. Secondary Outcome: Change From Baseline in Striatal Binding Ratio (SBR) in the Putamen as Measured by Single-Photon Emission Computed Tomography (SPECT) Imaging of the Dopamine Transporter (DaT) at Week 52
Description: SBR in the putamen as measured by SPECT imaging of the dopamine transporter (DaT) with 123^I-ioflupane (DaTscan™). The mean values reported are the adjusted mean values.
Time Frame: Baseline, Week 52
Population: The pharmacodynamic population was defined as a subset of the ITT population with at least 1 post-baseline pharmacodynamic measurement.
Measure: Mean (Standard Error); unit: striatal binding ratio
Arm/Group | PC Period: Placebo | PC Period: BIIB054 250 mg (Early Start) | PC Period: BIIB054 1250 mg (Early Start) | PC Period: BIIB054 3500 mg (Early Start)
Number analyzed (Participants) | 91 | 52 | 97 | 84
striatal binding ratio | -0.093 (0.0151) | -0.098 (0.0199) | -0.102 (0.0146) | -0.125 (0.0155)
Statistical Analysis 1: Comparison: PC Period: Placebo vs PC Period: BIIB054 250 mg (Early Start); Test type: Superiority — Adjusted mean, difference with placebo, 95% CI, and p-value were based on an MMRM model, with change from baseline in DaT/SPECT parameter as dependent variable and with fixed effects of treatment group, region, time, treatment group-by-time interaction, baseline MDS-UPDRS part I+II+III total score, baseline MDS-UPDRS part I+II+III total score by time interaction, baseline DaT/SPECT values and baseline DaT/SPECT by time interaction; p = 0.8274, Mixed Model for Repeated Measures; Difference = -0.005, 95% CI 2-sided [-0.0548 to 0.0438]
Statistical Analysis 2: Comparison: PC Period: Placebo vs PC Period: BIIB054 1250 mg (Early Start); Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.6671, Mixed Model for Repeated Measures; Difference = -0.009, 95% CI 2-sided [-0.0504 to 0.0323]
Statistical Analysis 3: Comparison: PC Period: Placebo vs PC Period: BIIB054 3500 mg (Early Start); Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.1313, Mixed Model for Repeated Measures; Difference = -0.033, 95% CI 2-sided [-0.0751 to 0.0098]

13. Secondary Outcome: Change From Baseline in SBR in the Striatum as Measured by SPECT Imaging of the DaT at Week 52
Description: SBR in the striatum as measured by SPECT imaging of the DaT with 123^I-ioflupane (DaTscan™). The mean values reported are the adjusted mean values.
Time Frame: Baseline, Week 52
Population: as for outcome 12
Measure: Mean (Standard Error); unit: striatal binding ratio
Arm/Group | PC Period: Placebo | PC Period: BIIB054 250 mg (Early Start) | PC Period: BIIB054 1250 mg (Early Start) | PC Period: BIIB054 3500 mg (Early Start)
Number analyzed (Participants) | 91 | 52 | 97 | 84
striatal binding ratio | -0.081 (0.0145) | -0.090 (0.0191) | -0.081 (0.0140) | -0.108 (0.0148)
Statistical Analysis 1: Comparison: PC Period: Placebo vs PC Period: BIIB054 250 mg (Early Start); Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.7079, Mixed Model for Repeated Measures; Difference = -0.009, 95% CI 2-sided [-0.0562 to 0.0382]
Statistical Analysis 2: Comparison: PC Period: Placebo vs PC Period: BIIB054 1250 mg (Early Start); Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.9835, Mixed Model for Repeated Measures; Difference = -0.000, 95% CI 2-sided [-0.0400 to 0.0392]
Statistical Analysis 3: Comparison: PC Period: Placebo vs PC Period: BIIB054 3500 mg (Early Start); Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.1869, Mixed Model for Repeated Measures; Difference = -0.027, 95% CI 2-sided [-0.0682 to 0.0134]

14. Secondary Outcome: Change From Baseline in SBR in the Caudate as Measured by SPECT Imaging of the DaT at Week 52
Description: SBR in the caudate as measured by SPECT imaging of the DaT with 123^I-ioflupane (DaTscan™). The mean values reported are the adjusted mean values.
Time Frame: Baseline, Week 52
Population: as for outcome 12
Measure: Mean (Standard Error); unit: striatal binding ratio
Arm/Group | PC Period: Placebo | PC Period: BIIB054 250 mg (Early Start) | PC Period: BIIB054 1250 mg (Early Start) | PC Period: BIIB054 3500 mg (Early Start)
Number analyzed (Participants) | 91 | 52 | 97 | 84
striatal binding ratio | -0.067 (0.0166) | -0.075 (0.0219) | -0.060 (0.0161) | -0.089 (0.0171)
Statistical Analysis 1: Comparison: PC Period: Placebo vs PC Period: BIIB054 250 mg (Early Start); Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.7585, Mixed Model for Repeated Measures; Difference = -0.008, 95% CI 2-sided [-0.0625 to 0.0456]
Statistical Analysis 2: Comparison: PC Period: Placebo vs PC Period: BIIB054 1250 mg (Early Start); Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.7808, Mixed Model for Repeated Measures; Difference = 0.006, 95% CI 2-sided [-0.0391 to 0.0520]
Statistical Analysis 3: Comparison: PC Period: Placebo vs PC Period: BIIB054 3500 mg (Early Start); Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.3532, Mixed Model for Repeated Measures; Difference = -0.022, 95% CI 2-sided [-0.0691 to 0.0248]

15. Secondary Outcome: Percentage of Participants With Anti-BIIB054 Antibodies in the Serum
Time Frame: Up to Week 144
Population: The analysis population for immunogenicity was defined as all participants in the safety population. As prespecified in the protocol, the data for the delayed start BIIB054 were pooled from Placebo/BIIB054 250/1250/3500 mg for the analysis of this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | PC Period: Placebo to BIIB054 250 mg/ 1250 mg / 3500 mg (Delayed Start - Pooled) | PC Period: Early Start BIIB054 250 mg | PC Period: Early Start BIIB054 1250 mg | PC Period: Early Start BIIB054 3500 mg
Number analyzed (Participants) | 96 | 55 | 100 | 99
percentage of participants | 0 | 1.8 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Safety Population included all participants who received at least one dose of the study treatment (BIIB054 250 mg, 1250 mg, 3500 mg).
Arm/Group | PC Period: Placebo | PC Period: BIIB054 250 mg (Early Start) | PC Period: BIIB054 1250 mg (Early Start) | PC Period: BIIB054 3500 mg (Early Start) | DBE Period: Placebo to BIIB054 250 mg (Delayed Start) | DBE Period: Placebo to BIIB054 1250 mg (Delayed Start) | DBE Period: Placebo to BIIB054 3500 mg (Delayed Start) | DBE Period: BIIB054 250 mg (Early Start) | DBE Period: BIIB054 1250 mg (Early Start) | DBE Period: BIIB054 3500 mg (Early Start)
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/55 | 0/102 | 0/100 | 0/20 | 0/37 | 0/39 | 0/52 | 0/100 | 1/94
Serious Adverse Events (participants affected / at risk) | 7/100 | 4/55 | 4/102 | 6/100 | 2/20 | 3/37 | 3/39 | 3/52 | 5/100 | 7/94
Other Adverse Events (participants affected / at risk) | 58/100 | 32/55 | 61/102 | 63/100 | 16/20 | 22/37 | 22/39 | 25/52 | 51/100 | 56/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PC Period: Placebo (N=100) | PC Period: BIIB054 250 mg (Early Start) (N=55) | PC Period: BIIB054 1250 mg (Early Start) (N=102) | PC Period: BIIB054 3500 mg (Early Start) (N=100) | DBE Period: Placebo to BIIB054 250 mg (Delayed Start) (N=20) | DBE Period: Placebo to BIIB054 1250 mg (Delayed Start) (N=37) | DBE Period: Placebo to BIIB054 3500 mg (Delayed Start) (N=39) | DBE Period: BIIB054 250 mg (Early Start) (N=52) | DBE Period: BIIB054 1250 mg (Early Start) (N=100) | DBE Period: BIIB054 3500 mg (Early Start) (N=94)
Monoclonal B-cell lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intracranial mass (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PC Period: Placebo (N=100) | PC Period: BIIB054 250 mg (Early Start) (N=55) | PC Period: BIIB054 1250 mg (Early Start) (N=102) | PC Period: BIIB054 3500 mg (Early Start) (N=100) | DBE Period: Placebo to BIIB054 250 mg (Delayed Start) (N=20) | DBE Period: Placebo to BIIB054 1250 mg (Delayed Start) (N=37) | DBE Period: Placebo to BIIB054 3500 mg (Delayed Start) (N=39) | DBE Period: BIIB054 250 mg (Early Start) (N=52) | DBE Period: BIIB054 1250 mg (Early Start) (N=100) | DBE Period: BIIB054 3500 mg (Early Start) (N=94)
Constipation (Gastrointestinal disorders) | 5 | 3 | 5 | 6 | 1 | 2 | 1 | 1 | 4 | 7
Diarrhoea (Gastrointestinal disorders) | 4 | 5 | 5 | 6 | 1 | 0 | 0 | 1 | 2 | 3
Nausea (Gastrointestinal disorders) | 6 | 1 | 6 | 6 | 1 | 2 | 4 | 2 | 4 | 7
Fatigue (General disorders) | 5 | 2 | 3 | 9 | 1 | 0 | 0 | 1 | 4 | 5
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 6 | 3
Influenza (Infections and infestations) | 3 | 1 | 7 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 12 | 10 | 10 | 13 | 2 | 0 | 0 | 2 | 4 | 5
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 6 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 3 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 5 | 5 | 6 | 14 | 2 | 2 | 3 | 10 | 16 | 16
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 5 | 9 | 11 | 1 | 4 | 3 | 3 | 7 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 3 | 8 | 13 | 0 | 4 | 6 | 5 | 5 | 8
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4 | 5 | 1 | 0 | 1 | 2 | 2 | 2 | 2
Dizziness (Nervous system disorders) | 3 | 4 | 9 | 6 | 0 | 2 | 2 | 1 | 4 | 4
Headache (Nervous system disorders) | 18 | 6 | 19 | 21 | 3 | 5 | 5 | 1 | 7 | 12
Parkinson's disease (Nervous system disorders) | 1 | 4 | 9 | 8 | 1 | 1 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 4 | 0 | 9 | 5 | 1 | 1 | 2 | 1 | 1 | 4
Depression (Psychiatric disorders) | 1 | 3 | 3 | 3 | 1 | 2 | 0 | 0 | 2 | 4
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 3 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 5 | 0 | 0 | 3 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 5 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia ear (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Calcium deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study did not meet its primary outcome measure for year 1 and did not demonstrate efficacy on key secondary outcome measures; additional pre-specified analyses at week 72 confirmed the study did not provide evidence of efficacy; resulting in the development of BIIB054 for Parkinson's disease to be discontinued and SPARK study was closed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT03318523/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT03318523/SAP_001.pdf